CLINICAL TRIAL: NCT02216292
Title: Impact of Preterm Single Donor Milk on Enteral Feeding in Very Low Birth Weight Infants
Brief Title: Impact of Preterm Single Donor Milk in Very Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, MD, Assoc. Prof., Medical University of Vienna
Other Study IDs: PSDM001
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Infant, Premature, Diseases
Keywords: preterm single donor milk; human milk; very lo birth weight infants; enteral feedings; NEC
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm Single Donor Milk Group: The prospective study group = preterm single donor milk group (PSDM-Group) from June 2012 - April 2013
  Interventions: Other: Preterm Single Donor Milk Group
- Control Group: Retrospective control group receiving no donor milk = control group from March 2011 - May 2012
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Control Group — Infants received preterm formula during their first days of life until breastmilk from their own mother was available
  Groups: Control Group
Other: Preterm Single Donor Milk Group — Infants received preterm single donor milk during their first days of life until breastmilk from their own mother was available
  Groups: Preterm Single Donor Milk Group

SUMMARY:
Human milk is the best source of enteral nutrition for the preterm infant. However during the infants first hours and days of life breastmilk from the own mother is usually not available. Until May 2012 the practice in the Neonatal Division of the Department of Pediatrics /Medical University Vienna was to start with formula feedings within the first 6 hours of life of a premature infant and switch over to breastmilk as soon it was available. In June 2012 the investigators changed this feeding regimen and started to use single donor milk of mothers of preterm infants for the first hours and days of the preterm infants life. In a prospective observational study the investigators evaluated the impact of single donor milk from preterm infants on time to full enteral feedings, gastrointestinal tolerance and NEC incidence in preterm infants with a birthweight below 1500 grams and a gestational below 32 weeks. Data will be compared with a historical control group starting with preterm formula as source of enteral nutrition. The investigators hypothesize that starting enteral nutrition with single donor milk of mothers from preterm infants with shorten time to full enteral feedings.

ELIGIBILITY:
Inclusion Criteria:

* very low birth weight infants with a birthweight <1500g
* Gestational Age <32 weeks
* Informed consent

Exclusion Criteria:

* major congenital malformations
* systemic metabolic diseases
* short bowl syndrome
* gastrointestinal abnormalities
* when preterm infant was transferred or discharged

Ages: 1 Minute to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: inborn very low birth weight infants with a birthweight <1500g and a gestational age <32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to full enteral feeding | birth up to 40 weeks of gestation
  Full enteral feedings are defined as an enteral inane of 135-145ml/kg/d

SECONDARY OUTCOMES:
necrotizing enterocolitis | birth to 40 weeks of gestation
  Necrotising enterocolitis (NEC) was defined according to the stages by Bell as proven NEC grade 2a.
Gastric residuals | birth to 7th day of life
  Gastric residuals are a parameter for gastrointestinal tolerance and are determined every three hours before the next meal is given and are aspirated via a gastric tube Gastric residuals are measured in ml/kg per meal. Furthermore the color is documented (milky, clear, mucous, bile stained, bloody)
Frequency of stool | birth until 14th day of life
  Number of stools per day
culture positive sepsis | birth to 40th week of gestation

OTHER OUTCOMES:
body weight | birth to 40th week of gestation
  body weight in gram is measured every second day.

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, Prof.MD, Principal Investigator — Medical University of Vienna, Department of Pediatrics
Locations (1):
- Medical University of Vienna, Vienna, Austria